CLINICAL TRIAL: NCT06102213
Title: A Randomized, Open-Label, Multicenter, Phase 2a Study To Evaluate The Safety And Efficacy of PBCLN-010 In Combination With PBCLN-014 in Participants Receiving Allogeneic Hematopoietic Cell Transplantation (Allo-HCT)
Brief Title: Study To Evaluate The Safety And Efficacy of PBCLN-010 In Combination With PBCLN-014 in Participants Receiving Allogeneic Hematopoietic Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision to terminate the study early
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-CT-001
Record Dates: First submitted 2023-10-09; First posted 2023-10-26 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-10

CONDITIONS: Hematologic Malignancy
Keywords: allo-hct; microbiome; gut engraftment
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Health Maintenance Organizations

STUDY DESIGN:
Intervention Model Description: 3 cohorts: Cohort A and B receive combination study drug in difference doses (Cohort A receives HMO 9.0 g and B. infantis; Cohort B received HMO 4.5 g and B. infantis) Cohort C does not receive study drug
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: HMO 9.0 g and B. infantis (Experimental): HMO will be administered at 9.0 g orally twice a day (BID), and B. infantis will be administered orally twice a day (BID) (total of 43 days of dosing).
  Interventions: Drug: B. infantis (PBCLN-014) and Human Milk Oligosaccharides (HMO) (PBCLN-010)
- Cohort B: HMO 4.5 g and B. infantis (Experimental): HMO will be administered at 4.5 g orally BID, and B. infantis will be administered orally BID (total of 43 days of dosing).
  Interventions: Drug: B. infantis (PBCLN-014) and Human Milk Oligosaccharides (HMO) (PBCLN-010)
- Cohort C (No Intervention): Participants in this cohort will not receive any study drug

INTERVENTIONS:
Drug: B. infantis (PBCLN-014) and Human Milk Oligosaccharides (HMO) (PBCLN-010) — PBCLN-010: Human Milk Oligosaccharides (HMO). PBCLN-014: B. infantis.
  Arms: Cohort A: HMO 9.0 g and B. infantis; Cohort B: HMO 4.5 g and B. infantis

SUMMARY:
This is a Phase 2a, open-label, multicenter study to evaluate the safety and efficacy of HMO (PBCLN-010) and B. infantis (PBCLN-014) on the gut microbiome and GI domination by pathobionts in participants receiving allo-HCT.

Approximately 60 participants will be enrolled in this study, and all participants will undergo screening assessments up to 28 days before the first study drug dose (D 7). Participants meeting all the eligibility criteria based on the screening assessments will be enrolled and randomly assigned to 1 of the 3 cohorts:

* Cohort A (HMO 9.0 g and B. infantis) BID
* Cohort B (HMO 4.5 g and B. infantis) BID
* Cohort C (Control Cohort): Participants in this cohort will not receive any study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-specific procedure or treatment.
2. Male and female participants 18 to 75 years of age at the time of informed consent.
3. Planning to receive a first allo-HCT.
4. Able to comply with protocol requirements.

Exclusion Criteria:

1. Participants with prior bowel resection resulting in colostomy
2. Serious medical or psychiatric illness likely to interfere with participation in study.
3. History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions.
4. Female participants who are pregnant, breastfeeding, lactating, or planning to become pregnant during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of safety and tolerability measures assessed through adverse events, serious adverse events, and adverse events of special interest per treatment group | before treatment, during treatment, or ≤ 56 days after cessation of treatment
Rate of gut engraftment of B. infantis through Day 180 among recipients of PBCLN-010 in combination with PBCLN-014 compared with standard of care (SOC) (control cohort). | Through study completion,180 days
Duration of gut engraftment of B. infantis through Day 180 among recipients of PBCLN-010 in combination with PBCLN-014 compared with standard of care (SOC) (control cohort). | Through study completion,180 days

SECONDARY OUTCOMES:
Measures of safety and tolerability by physical examinations examined by cohort to assess the effect of oral administration of PBCLN-010 in combination with PBCLN-014 | Dosing period, 43 days
Measuring the incidence of bloodstream infections, use of anti-infective agents, frequency/length of hospitalizations stays to evaluate the incidence of the infection and other safety events among recipients of study drug compared with SOC | Through study completion,180 days
Measuring temperature ≥ 38.0°C (100.4°F) sustained over a 1-hour period concurrent with ANC < 500 cells/mm3 to determine the incidence and duration of febrile neutropenia | Day -7 through neutrophil engraftment
Measuring cases of acute graft versus host disease (aGvHD) to determine the cumulative incidence or rate of acute graft versus host disease (aGvHD) at D180 | Through study completion,180 days

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Time Frame: To be determined
Access Criteria: To be determined